CLINICAL TRIAL: NCT06673199
Title: The Influence of the Japanese "washoku" Diet on the Composition of the Gut Microbiota and Its Metabolites in Overweight or Obese Postmenopausal Women
Brief Title: The Influence of the "washoku" Diet on the Gut Microbiota in Postmenopausal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joanna Bajerska (Other)
Responsible Party: Sponsor-Investigator, Joanna Bajerska, Associate Professor, Poznan University of Life Sciences
Organization: Poznan University of Life Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 661/24-Washoku diet
Record Dates: First submitted 2024-10-29; First posted 2024-11-04 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Menopause
Keywords: menopause; microbiota; isoflavones

STUDY DESIGN:
Intervention Model Description: Postmenopausal women (n=40), aged 45-65.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Washoku diet (Experimental): Participants assigned to the washoku group will be introduced to the principles of a healthy eating plate, which will be supplemented with elements of the washoku diet (30 g of roasted black soybeans and 5 g of wakame).
  Interventions: Dietary Supplement: Washoku diet
- Control group (No Intervention): Participants assigned to the control group will receive only dietary recommendations consistent with the healthy eating plate.

INTERVENTIONS:
Dietary Supplement: Washoku diet — The Washoku diet will consist of following the principles of a healthy eating plate, which will be supplemented with elements of the Washoku diet (30g of roasted black soybeans and 5g of wakame). Food products will be given to women on the day of the first meeting. The Washoku diet will be used for 7 days a week for a period of 1 month (4 weeks).
  Arms: Washoku diet

SUMMARY:
Menopause is a special period in a woman's life, when a sudden drop in estrogen levels leads to the cessation of menstrual cycles. Hormonal changes and a decreasing metabolic rate contribute to weight gain and the appearance of numerous metabolic disorders, such as dyslipidemia, impaired glucose tolerance, insulin resistance, hyperinsulinemia, and type 2 diabetes. Currently, effective and inexpensive dietary therapeutic solutions are being sought to improve the health of this group of women. It is suggested that the Japanese washoku diet, which includes products rich in isoflavones, fiber (soy products) and unsaturated omega-3 fatty acids (fish, seaweed), may be a good solution, as it contributes to the regulation of hormonal balance, lowering cholesterol levels, and reducing the risk of insulin resistance. Moreover, the composition of such a diet may also affect the diversity of the intestinal microbiota and the production of its metabolites, such as short-chain fatty acids, and thus contribute to the improvement of patients' health. Taking the above into account, the aim of the study will be to assess the effect of the Japanese washoku diet on the composition of the intestinal microbiota and its metabolites in a group of overweight or obese women after natural menopause.

Specific objectives:

* Assessment of anthropometric parameters (body weight, height, waist circumference, hip circumference) and body composition and bone density.
* Assessment of parameters of carbohydrate metabolism (glucose, insulin concentration), lipid metabolism (total cholesterol (T-C), low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C), non-HDL cholesterol (non-HDL-C) and triglycerides).
* Analysis of intestinal microbiota, short-chain fatty acids in the feces of women.

DETAILED DESCRIPTION:
Women who meet the criteria for inclusion in the study for a period of 4 weeks will be randomly assigned to one of two groups: 1. The intervention group will follow the principles of the healthy eating plate, which will be supplemented with elements of the washoku diet (30 g of roasted black soybeans and 5 g of wakame); 2. The control group will be covered only by the principles of the healthy eating plate.

All participants will receive a brochure with information on the recommended portion sizes of individual product groups in the daily diet, recipes for dishes based on roasted black soybeans and wakame. Before and after the study, in addition to anthropometric measurements (body weight, waist circumference, hip circumference), body composition and bone mineral density, an assessment of the diet (using a semi-quantitative questionnaire of food frequency, as well as the current recording method from the last 4 days) and the level of physical activity will be carried out. Additionally, the women will be asked to collect a daily portion of urine to assess the concentration of soy isoflavones and to determine the content of sodium, potassium and magnesium. Women will also have their blood (18 ml) collected to assess selected biochemical parameters (glucose, insulin, total cholesterol (TC), low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C), non-HDL cholesterol (non-HDL-C) and triglycerides). A stool sample will also be collected to assess the composition of the intestinal microbiota and its metabolites, i.e. short-chain fatty acids. Recruitment will take place via social networking sites, i.e. Facebook.

The following specific analyses were planned:

* Assessment of anthropometric parameters (height, body weight, hips and waist circumference)
* Analysis of body composition and bone mineral density
* Assessment of nutritional status (selected metabolic parameters such as glucose metabolism (glucose, insulin concentration), lipid metabolism (total cholesterol (T-C), LDL cholesterol (LDL-C), HDL cholesterol (HDL-C), non-HDL cholesterol (non-HDL-C) and triglycerides).
* Assessment of dietary habits (a semi-quantitative questionnaire on the frequency of food intake, additionally supplemented by the current recording method from the last 4 days.)
* Assessment of intestinal microbiota composition
* Assessment of fecal short-chain fatty acid concentration
* Assessment of urine soy isoflavones concentration

Normality of the obtained data distribution will be tested using the Shapiro-Wilk test. The Kruskal-Wallis test then will be used for nonnormally distributed data and the Tukey HSD test will be used for normally distributed data. A p value of less than 0.05 was considered statistically. The microbiota composition will be analyzed using RStudio (R version 4.0.3 (2020-10-10)) with packages including phyloseq, microbiome, and vegan. Taxa will be filtered by removing all those not assigned to any phylum. Only taxa with abundances over 0.25% in at least one sample will left in the dataset. All analyses of gut microbiota composition will be performed on the basis of the relative abundances (RA) of the OTUs (Operational Taxonomic Units).

The data collected in the planned studies will include the results of measurements and their statistical analyzes. All data will be collected directly by team members and coded. Detailed instructions on data collection will be prepared by the team leader and each member will need to read and receive appropriate training. All biochemical and anthropometric measurements will be performed in at least two repetitions and will be checked by another team member. All used specialized equipment will be properly calibrated before each use (scale, body composition analyzer, Nanodrop spectrophotometer).

ELIGIBILITY:
Inclusion Criteria:

* age 45 to 65,
* at least one year after natural menopause,
* BMI > 25 kg/m2
* waist circumference > 80 cm.

Exclusion Criteria:

* use of hormone replacement therapy;
* taking antibiotics or probiotics in the last 6 months from the date of commencement of the scientific experiment,
* taking medications regulating carbohydrate or lipid metabolism in the last 4 weeks from the date of commencement of the scientific experiment,
* taking medications regulating body weight in the last 3 months from the date of commencement of the scientific experiment,
* diseases of the thyroid gland, liver, heart, kidneys, digestive system, anemia, neoplastic diseases,
* smoking or alcohol consumption in amounts exceeding 100 g/week.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-16 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-11-12 (Estimated)

PRIMARY OUTCOMES:
Change in composition of the intestinal microbiota | Week 0 (pre-intervention) and week 4 (post-intervention)
  Participants will be asked to provide stool samples at each scheduled meeting. Detailed instructions on sample collection and transport will be provided by the people conducting the study, and participants will receive containers containing preservative liquid. Bacterial DNA will be isolated from the provided stool samples using the QIAmp Fast DNA Stool Mini Kit. Then, the DNA will be properly secured and sent to an external company, Genomed S.A. (Warsaw, Poland), in which the assessment of microbiota will be carried out by metagenomic 16s rRNA sequencing using the V3-V4 region. Then, a bioinformatics analysis will be performed in the R environment using packages such as phyloseq, vegan, microbiome.
Change in body weight | Week 0 (pre-intervention) and week 4 (post-intervention)
  Body weight measurement in a standing position, without shoes, in light clothing, on an electronic scale with an accuracy of 0.1 kg.
Change in body composition | Week 0 (pre-intervention), week 4, week 8 and week 12 (post-intervention)
  Body composition will be measured using dual-energy X-ray absorptiometry (DXA) as a method that uses the phenomenon of weakening the beam of ionizing radiation passing through tissues of various densities. This method is safe and non-invasive. The mass of adipose tissue, including visceral fat tissue, the mass of lean tissue are measured. (expressed in the same unit - kilograms)
Change in circumferences | Week 0 (pre-intervention) and week 4 (post-intervention)
  Waist and hip measurements will be taken using an elastic tape. Waist circumference measurement - the tape is placed horizontally or slightly obliquely halfway between the lower edge of the ribs and the upper crest of the ilium. Measurement performed during apnea.
Change in lipid profile | Week 0 (pre-intervention) and week 4 (post-intervention)
  Blood will be collected four times from the antecubital vein on an empty stomach, into test tubes with clotting granules (a single sample will amount to a total of 18 ml). The serum will be obtained by centrifugation of a venous blood clot. Total cholesterol (T-C), low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C) and triglycerides concentrations will be determined by a certified external laboratory. The nonHDL-C parameter will be calculated using the formula: nonHDL-C = T-C - HDL-C. (expressed in the same unit - mg/dl or mmol/l).
Change in glucose metabolism | Week 0 (pre-intervention) and week 4 (post-intervention)
  Blood will be collected four times from the antecubital vein on an empty stomach, into test tubes with clotting granules (a single sample will amount to a total of 18 ml). The serum will be obtained by centrifugation of a venous blood clot. Insulin concentration will be performed using the ELISA enzyme-linked immunosorbent assay, while glucose will be determined by a certified external laboratory. (expressed in the same unit - mg/dl or mmol/l).
Change in urinary isoflavone content | Week 0 (pre-intervention) and week 4 (post-intervention)
  Soy isoflavone concentrations will be assessed in a 24-hour urine sample provided by women before and after the study using high-performance liquid chromatography.
Change in urine pH | Week 0 (pre-intervention) and week 4 (post-intervention)
  pH will be assessed in a 24-hour urine sample provided by women before and after the study using litmus paper or laboratory pH meter.
Change in urine creatinine | Week 0 (pre-intervention) and week 4 (post-intervention)
  Creatinine concentration will be assessed in a 24-hour urine sample provided by women before and after the study using high-performance liquid chromatography.
Change in urine sodium and magnesium | Week 0 (pre-intervention) and week 4 (post-intervention)
  Sodium and magnesium concentrations will be assessed in a 24-hour urine sample provided by women before and after the study using automatic electrolyte analyzer.

SECONDARY OUTCOMES:
Changes in results of nutrition assessment | Week 0 (pre-intervention) and week 4 (post-intervention)
  Nutrition assessment will be carried out using food frequency questionnaire (FFQ) which concerns the frequency of consumption of 62 food groups in the last 12 months. The obtained data (frequency of food consumption rated from 1 to 6) will then be transformed into semi-quantitative data by ranking - assigning values 0-2 to the categories of food consumption frequency. Then diet quality indicators will be calculated - pro-Healthy-Diet-Index-10 (pHDI - range 0-20), non-Healthy-Diet-Index-14 (nHDI - range 0 - 28), Diet-Quality-Index (DQI - range -100-100). The higher the value of the pHDI or DQI index, the greater the intensity of nutritional features beneficial to health and the better the quality of the diet. The higher the value of the nHDI index, the greater the intensity of nutritional characteristics unfavorable for health and the worse the quality of the diet. In addition, this method will be supplemented with the current dietary recording for the last 4 days.
Change in bone density | Week 0 (pre-intervention) and week 4 (post-intervention)
  Bone density will be measured using dual-energy X-ray absorptiometry (DXA) as a method that uses the phenomenon of weakening the beam of ionizing radiation passing through tissues of various densities. This method is safe and non-invasive.
Change in the concentration of short-chain fatty acids in feces | Week 0 (pre-intervention) and week 4 (post-intervention)
  Quantitative and qualitative determination of short-chain fatty acids in feces will be carried out using the gas chromatography method with flame ionization detection (GC-FID). The research will be carried out at the Department and Department of Bromatology, Medical University of Poznań.
Change in intestinal barrier integrity | Week 0 (pre-intervention) and week 4 (post-intervention)
  Blood will be collected four times from the antecubital vein on an empty stomach, into test tubes with clotting granules (a single sample will amount to a total of 18 ml). The serum will be obtained by centrifugation of a venous blood clot. Lipopolysaccharide concentrations will be assessed using the ELISA enzyme-linked immunosorbent assay.

CONTACTS AND LOCATIONS:
Overall Officials: Agata Chmurzyńska, Prof., Study Chair — Department of Human Nutrition and Dietetics, Poznań University of Life Sciences
Locations (1):
- Poznań University of Life Sciences, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Yes
Numerical data, statistics and graphs data will be deposited in the Open Data Repository RepOD - the PULS institutional repository, and made publicly available in the Repository at the latest at the time when the publication presenting research data is published including a maximum 36-month embargo period due to the requirements and specifics of the publication of the article presenting the research results. Upon publication, the embargo will be lifted immediately.
  Unless there is a clear indication to the contrary, the data will be made available in the RepOD repository under a CC BY 4.0 license.
  Raw and processed data will be stored for at least 10 years. Personal data will be deleted after the pseudonymization process.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD data will be made available after publication of all planned articles presenting the results of the planned experiment for a period of 10 years.
Access Criteria: All persons having access to data have to be authorised to process personal data. A secured work e-mail is used for correspondence. Access to collected and processed sensitive data will be limited solely to the group of authorised users. The Head of the project authorises individuals to have access to data.
  The e-mail requesting access to the IPD should include your name and surname, academic degree and affiliation. Data will only be made available after the person's identity has been verified and the purpose of using the data is clear (e.g. meta-analysis). Then, the data owner will verify the need to have the data and send it in a password-protected form. All data will be pseudonymized.

REFERENCES:
- [Background] Yang M, Wen S, Zhang J, Peng J, Shen X, Xu L. Systematic Review and Meta-analysis: Changes of Gut Microbiota before and after Menopause. Dis Markers. 2022 Jul 25;2022:3767373. doi: 10.1155/2022/3767373. eCollection 2022. PMID 35923245
- [Background] Kanai T, Matsuoka K, Naganuma M, Hayashi A, Hisamatsu T. Diet, microbiota, and inflammatory bowel disease: lessons from Japanese foods. Korean J Intern Med. 2014 Jul;29(4):409-15. doi: 10.3904/kjim.2014.29.4.409. Epub 2014 Jun 27. PMID 25045286
- [Background] Seura T, Fukuwatari T. Japanese Diet Score Is Associated with Gut Microbiota Composition in Young Japanese Adults. J Nutr Sci Vitaminol (Tokyo). 2019;65(5):414-420. doi: 10.3177/jnsv.65.414. PMID 31666478
- [Background] Gabriel AS, Ninomiya K, Uneyama H. The Role of the Japanese Traditional Diet in Healthy and Sustainable Dietary Patterns around the World. Nutrients. 2018 Feb 3;10(2):173. doi: 10.3390/nu10020173. PMID 29401650
- [Background] Takahashi TA, Johnson KM. Menopause. Med Clin North Am. 2015 May;99(3):521-34. doi: 10.1016/j.mcna.2015.01.006. PMID 25841598